CLINICAL TRIAL: NCT04960618
Title: Pembrolizumab in Combination With Gemcitabine for Previously Treated Mycosis Fungoides and Sézary Syndrome: Efficacy and Characterization of Immune Response
Brief Title: Pembrolizumab in Combination With Gemcitabine in People With Advanced Mycosis Fungoides or Sézary Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-242
Record Dates: First submitted 2021-06-25; First posted 2021-07-14 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Mycosis Fungoides; Mycosis Fungoides/Sezary Syndrome; Sezary Syndrome; Sézary; Advanced Mycosis Fungoides
Keywords: Advanced Mycosis Fungoides; Mycosis Fungoides; Sezary Syndrome; 21-242; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Mycosis Fungoides; Sezary Syndrome | interventions — Gemcitabine; pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with confirmed mycosis fungoides/Sezary syndrome (Experimental): Participants will have confirmed mycosis fungoides/Sezary syndrome, disease stage IB (defined as patches, plaque, or papules that involve 10% of the skin surface viscera) or higher.
  Interventions: Drug: Gemcitabine; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Gemcitabine — Participants will receive gemcitabine 1000 mg/m2 on days 1 and 8 on 21-days cycles for up to 6 cycles
Drug: Pembrolizumab — Pembrolizumab 200 mg will be introduced with cycle 2 and will be given on day 1 of each 21-day cycle for up to 35 cycles

SUMMARY:
The purpose of this study is to find out whether the combination of pembrolizumab and gemcitabine is an effective treatment for mycosis fungoides and Sézary syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed mycosis fungoides/Sezary syndrome, disease stage IB (defined as patches, plaque, or papules that involve 10% of the skin surface viscera) or higher.
* Age ≥ 18 years.
* ECOG Performance Score between 0-1
* Receipt of at least one prior systemic therapy for MF/SS.
* Previous systemic anti-cancer therapy must have been discontinued at least 2 weeks prior to treatment. See section 6.2 Subject Exclusion Criteria for guidelines regarding adjuvant and maintenance therapy for prior malignancy.
* Topical or systemic steroids (equivalent to ≤ 10 mg/day of prednisone) may be considered if dose has been constant and discontinuation may lead to rebound flare in disease, adrenal insufficiency, and/or unnecessary suffering.
* Prior therapy with gemcitabine allowed.
* Refer to Table 1 for laboratory inclusion criteria.
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) as defined in Appendix C
  * A WOCBP who agrees to follow the contraceptive guidance in Appendix C
* A male participant must agree to use a contraception as detailed in Appendix C of this protocol from screening and through 6 months after the last dose of gemcitabine or 120 days after the last dose of pembrolizumab (whichever is later) and refrain from donating sperm during this period.

Table 1: Laboratory Parameters for Inclusion Criteria

System : Laboratory Value

Hematological Absolute neutrophil count (ANC): ≥ 1500/μL Platelets: ≥ 100 000/μL Hemoglobin: ≥ 9.0 g/dL or ≥ 5.6 mmol/L^a

Renal Creatinine OR Measured or calculated^b creatinine clearance (GFR can also be used in place of creatinine or CrCl): ≤ 1.5 × ULN OR ≥ 30 mL/min for participant with creatinine levels > 1.5 × institutional ULN

Hepatic Total bilirubin: ≤ 1.5 ×ULN OR direct bilirubin ≤ ULN for participants with total bilirubin levels >1.5 × ULN AST (SGOT) and ALT (SGPT): ≤ 2.5 × ULN (≤ 5 × ULN for participants with liver metastases)

Coagulation International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT): ≤ 1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants

ALT (SGPT)=alanine aminotransferase (serum glutamic pyruvic transaminase); AST (SGOT)=aspartate aminotransferase (serum glutamic oxaloacetic transaminase); GFR=glomerular filtration rate; ULN=upper limit of normal.

* a: Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.
* b: Creatinine clearance (CrCl) should be calculated per institutional standard.

Note: This table includes eligibility-defining laboratory value requirements for treatment; laboratory value requirements should be adapted according to local regulations and guidelines for the administration of specific chemotherapies.

Exclusion Criteria:

* A WOCBP who has a positive urine pregnancy test within 72 hours prior to the first dose of treatment (see Appendix C). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137).
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has an active infection requiring systemic therapy.
* Has a known additional malignancy that is progressing or has required active treatment within the past year. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention. A shorter timeframe down to 2 weeks may be acceptable if the investigator feels that this is in the best interests of the patient.
* Has received prior systemic anti-cancer therapy including investigational agents, phototherapy or radiotherapy within 4 weeks prior to the first dose of study intervention excluding topical steroids. A shorter timeframe down to 2 weeks may be acceptable if the investigator feels that this is in the best interests of the patient.
* Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤ 2 weeks of radiotherapy) to non-CNS disease.
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette- Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
* Has active autoimmune disease that has required systemic treatment in the past year (i.e. with use of disease modifying agents, corticosteroids (exceeding 10 mg daily of prednisone equivalent or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known active CNS lymphoma. Participants with previously treated CNS lymphoma may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
* Has severe hypersensitivity (≥ Grade 3) to pembrolizumab and/or any of its excipients.
* Adjuvant or maintenance therapy to reduce the risk of recurrence of other malignancy (other than T-cell lymphoma) is permissible after discussion with the Principal Investigator.
* Has a known history of Human Immunodeficiency Virus (HIV) infection.
* Has known active Hepatitis B (defined as Hepatitis B DNA detected by PCR) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Patients with evidence of prior hepatitis B infection require prophylaxis with entecavir or equivalent.
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Has had an allogenic tissue/solid organ transplant.
* Has a known history of active TB (Bacillus Tuberculosis).
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 6 months after the last dose of gemcitabine or 120 days after the last dose of pembrolizumab (whichever is later). See Appendix C for details regarding contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | 6 months
  Estimate overall response rate (ORR) using the composite global response criteria

CONTACTS AND LOCATIONS:
Overall Officials: Alison Moskowitz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All protocol activities), New York, New York
  - Columbia University, New York, New York
  - Memorial Sloan Kettering Nassau (Limited protocol activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org